CLINICAL TRIAL: NCT06747845
Title: ParpVax2: A Phase II Study Of Maintenance Niraparib Plus Ipilimumab In Patients With Metastatic Pancreatic Cancer Whose Disease Has Not Progressed On Platinum-Based Therapy
Brief Title: Maintenance Niraparib Plus Ipilimumab in Patients With Metastatic Pancreatic Adenocarcinoma Whose Disease Has Not Progressed on Platinum-Based Chemotherapy
Acronym: ParpVax2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Lustgarten Foundation (Other); GlaxoSmithKline (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19224
Record Dates: First submitted 2024-11-26; First posted 2024-12-24 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Adenocarcinoma Metastatic
Keywords: Niraparib; Ipilimumab; Pancreatic ductal adenocarcinoma; PDAC; Maintenance cancer therapy; Platinum-based therapy; PARP inhibitor; anti-CTLA-4 therapy
MeSH Terms: interventions — niraparib; IFL protocol; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Niraparib + Ipilimumab (Arm A) (Experimental): niraparib + ipilimumab
  Interventions: Drug: Niraparib; Drug: Ipilimumab
- FOLFIRI (Arm B) (Other): standard chemotherapy FOLFIRI
  Interventions: Drug: FOLFIRI

INTERVENTIONS:
Drug: Niraparib — Niraparib 200mg PO daily on days 1-21 of each 21-day cycle.
  Other Names: Arm A
  Arms: Niraparib + Ipilimumab (Arm A)
Drug: FOLFIRI — Standard chemotherapy FOLFIRI (5-fluorouracil, folinic acid, and irinotecan) will be administered intravenously every 14 days of a 28-day cycle.
  Other Names: Arm B
  Arms: FOLFIRI (Arm B)
Drug: Ipilimumab — Ipilimumab 3mg/kg IV day 1 of each cycle, for the first 4 cycles only.
  Other Names: Arm A
  Arms: Niraparib + Ipilimumab (Arm A)

SUMMARY:
The main goal of this study is to look at the effectiveness and anti-tumor activity (preventing growth of the tumor) of the drugs niraparib and ipilimumab, on the patients and their pancreatic cancer. This study will involve two different treatment arms. In Arm A, patients will receive niraparib plus ipilimumab. In Arm B, patients will receive standard chemotherapy.

The main questions the study aims to answer are:

* Does niraparib plus ipilimumab slow down tumor growth in patients with pancreatic cancer?
* What medical problems do participants have when taking niraparib plus ipilimumab?

Participants will:

* Undergo screening procedures to evaluate their cancer, overall health, and suitability for the study
* After passing screening, will be randomized to Arm A or B and be scheduled to receive niraparib plus ipilimumab (Arm A) or chemotherapy (Arm B)
* Receive niraparib plus ipilimumab every 3 weeks (Arm A)
* Receive chemotherapy every 2 weeks (Arm B)
* Visit the clinic for regular checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of pancreatic adenocarcinoma with metastatic disease
* ≥18 years of age
* Patients must be able to understand the study procedures and agree to participate in the study by providing written informed consent
* Participants must have received 8-12 cycles (4-6 months) of first-line FOLFIRINOX or modified FOLFIRINOX for metastatic disease with stable disease or better. Patients treated with liposomal irinotecan with oxaliplatin, 5-fluorouracil and leucovorin (NALIRIFOX) are also eligible. Patients who were initially treated with FOLFIRINOX or NALIRIFOX but stopped oxaliplatin because of toxicity are eligible for the trial.

  * Note: This requires at least stable imaging and a stable or decreasing tumor marker as applicable and as determined by the investigator.
* Measurable disease is not a requirement for study entry.

  * Note: The study will require that at least 80% of enrolled patients (ie 55 of all patients) are biopsiable at enrollment. The investigators may require measurable/biopsiable disease as the study progresses in order to achieve this goal.
* Participants must be willing to undergo a pre-treatment fresh tumor biopsy (if medically feasible).
* Participants must be willing to undergo an on-treatment tumor biopsy (if medically feasible).
* Female participant has a negative serum pregnancy test within 24 hours prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 6 months (females) or 30 days (males) after the last dose of study treatment, or is of nonchildbearing potential.
* Male patient agrees to use an adequate method of contraception starting with the first dose through 90 days after the last dose of study treatment.
* Adequate organ function confirmed by the following laboratory values obtained ≤7 days prior to the first day of study therapy:

  * Absolute neutrophil count (ANC) ≥1.5 x 109/L
  * Platelets>100 x 109/L
  * Hemoglobin ≥9g/dL
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x upper limit of normal (ULN); if liver metastases, then ≤5 x ULN
  * Total bilirubin ≤1.5 x ULN; if liver metastases or metabolic disorder such as Gilbert's syndrome, then ≤2.5 x ULN.
  * Serum creatinine ≤1.5 x ULN or estimated glomerular filtration rate (GFR) ≥45 mL/min using Cockcroft Gault formula.
* Eastern Cooperative Oncology (ECOG) performance status of 0 to 1.

Exclusion Criteria:

* Prior treatment with a PARP inhibitor, ipilimumab, or other cytotoxic T-lymphocyte-associated-4 protein (CTLA-4) inhibitor.
* Patients who have demonstrated resistance to FOLFIRINOX are not eligible to participate in this study
* Patients with known pathogenic/likely pathogenic germline or somatic alteration(s) in BRCA1, BRCA2, PALB2, RAD51C, or RAD51D.
* Patients with known mismatch repair deficiency or microsatellite instability-high cancer.
* Clinical evidence of uncontrolled malabsorption and/or any other gastrointestinal disorder or defect that would, in the opinion of the investigator, interfere with the absorption of niraparib
* Patients with uncontrolled hypertension, defined as systolic BP >140mmHg and/or diastolic BP >90mmHg
* Patients with a prior history of posterior reversible encephalopathy syndrome (PRES)
* Acute infection requiring intravenous antibiotics, intravenous antiviral or intravenous antifungal agents during the 14 days prior to first dose of study therapy
* Patients will be excluded if they have a history of or active autoimmune disease, defined as: patients with a history of inflammatory bowel disease are excluded from this study, as are patients with a history of symptomatic autoimmune disease (e.g. rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis e.g. Wegener's Granulomatosis); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome).

  * Note: Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Has a history of interstitial lung disease or active, non-infectious pneumonitis
* Has received a live vaccine within 4 weeks prior to the first dose of trial therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated and are allowed; however intranasal influenza vaccines (e.g. Flu-Mist®) are live attenuated vaccines and are not allowed.
* For fertile patient (female able to become pregnant or male able to father a child), refusal to use effective contraception during the period of the trial and:

  * Female patients refusing to use effective contraception for 6 months after the last dose of study drug.
  * Male patients refusing to use effective contraception for 90 days after the last dose of study drug.
* Received any systemic treatment for pancreatic cancer ≤14 days prior to first dose of therapy. Patients must not have had investigational therapy administered ≤ 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
* Patients will be excluded if they have a condition requiring systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses >10mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patient has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment.
* Non-study related minor surgical procedure ≤5 days, or major surgical procedure ≤21 days, prior to the first dose of therapy; in all cases, patients must be sufficiently recovered and stable before treatment administration.
* Active drug or alcohol use or dependence that would interfere with study compliance.
* Presence of any other condition that may increase the risk associated with study participation or may interfere with the interpretation of study results, and, in the opinion of the investigator, would make the patient inappropriate for entry into the study.
* Patient must not have any known history of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Patients must not be simultaneously enrolled in any therapeutic clinical trial
* Patients must not have had radiotherapy within 4 weeks of the first dose of study treatment
* Patients must not have a known hypersensitivity to the components of niraparib or the excipients
* Patients must not have received a transfusion (platelets or red blood cells) ≤ 4 weeks of the first dose of study treatment
* Patients must not be undergoing treatment for a second active cancer at the time of randomization. Exceptions include: (1) local therapies for skin cancers, (2) hormonal therapies for breast or prostate cancer without evidence of active disease. Patients may have a history of: (1) adequately treated nonmelanoma skin cancers, (2) curatively treated in situ cancer of the cervix, (3) curatively treated DCIS, (4) curatively treated stage I, grade 1 endometrial carcinoma, (5) other solid tumors and lymphomas (without bone marrow involvement) diagnosed at least five years prior to randomization and treated with no evidence of disease recurrence.
* Patients with active hepatitis B or hepatitis C infections, as defined by positive PCR testing, may not enroll.
* Patients with HIV may enroll, but must have an undetectable viral load at the time of enrollment and must be receiving a stable regimen of HAART.
* Patients must not have known, symptomatic brain or leptomeningeal metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-01-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in the experimental arm | From Cycle 1 (each cycle in Arm A is 21 days) Day 1 to disease progression, loss to follow-up or death from any cause, whichever came first, assessed up to 42 months.
  PFS is defined as the time from randomization to the occurrence of disease progression according to RECIST v1.1, as assessed by the investigator, or death from any cause. Median PFS and 95% confidence interval will be estimated from the Kaplan-Meier curve. In the primary outcome measure, PFS will be assessed in Arm A.

SECONDARY OUTCOMES:
Overall response rate (ORR) in the experimental arm | From first restaging assessment through completion of study treatment (maximum 42 months)
  The proportion of patients who achieve a complete or partial response, as determined by RECIST v1.1, in Arm A
Overall survival (OS) in the experimental arm | From Cycle 1 (each cycle in Arm A is 21 days) Day 1 until death, loss to follow-up, withdrawal of consent or until 5 years have passed, whichever occurs first
  Time from randomization to death from any cause in Arm A
Disease Control in the experimental arm | From Cycle 1 (each cycle in Arm A is 21 days) Day 1 to disease progression, loss to follow-up or death from any cause, whichever came first, assessed up to 42 months..
  Achieving stable disease (SD), partial response (PR), or complete response (CR) per RECIST v1.1, in Arm A
Safety and tolerability of Niraparib plus Ipilimumab in the experimental arm | From Cycle 1 (each cycle in Arm A is 21 days) Day 1 through 90 days after patient End of Treatment Visit
  The incidence of adverse events (AEs), clinical laboratory abnormalities and dose modifications, as determined by CTCAE v5.0, in Arm A
PFS in the control arm | From Cycle 1 (each cycle in Arm B is 28 days) Day 1 to disease progression, loss to follow-up or death from any cause, whichever came first, assessed up to 42 months.
  PFS is defined as the time from randomization to the occurrence of disease progression according to RECIST v1.1, as assessed by the investigator, or death from any cause. Median PFS and 95% confidence interval will be estimated from the Kaplan-Meier curve. In the secondary outcome measure, PFS will be assessed in Arm B.
OS in the control arm | From Cycle 1 (each cycle in Arm B is 28 days) Day 1 until death, loss to follow-up, withdrawal of consent or until 5 years have passed, whichever occurs first
  Time from randomization until death from any cause or last follow-up in Arm B
Overall response in evaluable patients within the control arm | From first restaging assessment through completion of study treatment (maximum 42 months)
  The proportion of patients who achieve a complete or partial response, as determined by RECIST v1.1, in Arm B

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/45/NCT06747845/Prot_SAP_000.pdf
  • Informed Consent Form (2025-01-21): https://cdn.clinicaltrials.gov/large-docs/45/NCT06747845/ICF_001.pdf